CLINICAL TRIAL: NCT04057703
Title: National Study Backed by a Rare Disease Cohort the Benefit / Risk Balance of Immunomodulatory Treatments Prescribed in the Child and Adolescent for Autoimmune Cytopenia.
Brief Title: Balance Benefit / Risk of Immunomodulatory Treatments at the Child and Adolescent for Autoimmune Cytopenia.
Acronym: VIGICAIRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHU BX 2013/24
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Immune Thrombocytopenic Purpura; Autoimmune Hemolytic Anemia; Evan Syndrome; Immunotherapy
Keywords: CEREVANCE; Pediatrics; Cohort
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune; Evans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In France, a national prospective cohort for monitoring children and adolescents with autoimmune cytopenia OBS'CEREVANCE is in place since 2004. It is coordinated in Bordeaux by the Center's team. Reference Rare Diseases CEREVANCE. It has been validated by the French Data Protection Authority in 2009 (information note and written consent). It had mid 2013 more of 900 patients, and the data collected make it possible to study intentionally to treat the therapeutic management of patients with Chronic Immune-Thrombocytopenic Purpura, from Autoimmune Hemolytic Anemia, or from EVANS syndrome.

This study evaluates efficacy and tolerance at 6 months of treatment immunomodulators prescribed in France in real conditions of use, in children and adolescents under the age of 18, for a Chronic Immune-Thrombocytopenic Purpura, an Autoimmune Hemolytic Anemia or a simultaneous EVANS syndrome.

DETAILED DESCRIPTION:
Chronic immunological thrombocytopenic purpura and anemia hemolytic autoimmune are rare autoimmune hematologic diseases, primary or secondary, affecting the child often very young, sometimes associated simultaneously or sequentially (Evans syndrome). They can be life-threatening, they in 20 to 50% of cases of prolonged dependence on immunosuppressants. The incidence of Immune-Thrombocytopenic Purpura is 2 to 5 / 100,000 inhabitants of under 18, the Autoimmune Hemolytic Anemia 5 to 10 times lower.

For the pediatric population, the experience reported in the literature is limited to individual cases or small series often retrospective and not comparative. It does not allow to have in 2013 a reasoning based on on evidence to define the second-line therapeutic strategy, in especially for Autoimmune Hemolytic Anemia where the therapeutic data are almost nonexistent. Splenectomy remains to this day the reference treatment of the Chronic Immune-Thrombocytopenic Purpura of the adult. In children, the therapeutic goal is to avoid it or to prevent it delay it. After failure of first-line treatments (immunoglobulins or corticosteroids) used for treatment of relapses or continuously, the main immunomodulatory treatments used in second line are azathioprine, ciclosporin, hydroxychloroquine, rituximab, mycophenolate mofetil, romiplostim, eltrombopag.

The benefit / risk balance of these 7 immunomodulatory treatments prescribed to the child for autoimmune cytopenia is presumed to be favorable based on the very limited data from the pediatric literature and the experience of most adults do not benefit from a specific marketing authorization.

ELIGIBILITY:
Inclusion Criteria:

* Patient initiating a first second-line immunomodulatory treatment (azathioprine, ciclosporine, eltrombopag, hydroxychloroquine, mycophénolate mofétil, rituximab, romiplostim), registered in the OBS'CEREVANCE database, presenting a Chronic Immune-Thrombocytopenic Purpura, Autoimmune Hemolytic Anemia or simultaneous EVANS syndrome.

Exclusion Criteria:

* Patient under immunosuppressant for another immunological pathology at the initiation of the first second line treatment,
* Patient treated with 2 second-line treatments on the same day,
* Oral refusal of participation of the patient or his legal representatives, after reading the information note specific for the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children or adolescents who have received one or more treatments of interest for a Chronic Immune-Thrombocytopenic Purpura, Autoimmune Hemolytic Anemia , or EVANS syndrome, in one of the 30 centers of the CEREVANCE network, will be identified and selected by the team CEREVANCE, in the OBS'CEREVANCE computer database created since 2004. The first second-line treatment they received will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2016-12-04 (Actual); Study Completion 2016-12-04 (Actual)

PRIMARY OUTCOMES:
Haemorrhagic sign - Grade ≥ 3 (Buchanan score) Presence of a haemorrhagic sign ≥grade 3 | At 6 months
  Presence of a haemorrhagic sign ≥ grade 3 = moderate bleeding (Buchanan score : from 0 to 5)
Thrombocytopenia Presence of thrombocytopenia <30 G / L | At 6 months
  Presence of thrombocytopenia <30 G / L
Need of a transfusion ? | At 6 months
  Performing a transfusion : yes or no ?
Immunoglobulin IV Immunoglobulin IV | At 6 months
  Immunoglobulin IV push
Corticoids push | At 6 months
  Corticoid push (no reduction of their number during treatment follow-up versus non-treatment period)
Need a splenectomy ? | At 6 months
  Performing a splenectomy : yes or no ?
Clinical signs of anemia | At 6 months
  Presence of clinical signs of anemia ≥ grade 2 = Subject bedridden less than 50% of the day (WHO score : from 0 to 4)
Anemia | At 6 months
  Presence of anemia <7g / dl
  Presence of anemia <7g / dl
Introduction of a new immunomodulatory treatment | At 6 months
  Introduction of a new immunomodulatory treatment : yes or no ?
Stop treatment or not ? | At 6 months
  Stop treatment because of failure, intolerance or non-compliance

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie ALADJIDI, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No
Through this program, a coordinated and centralized analysis of reliable pharmacovigilance data will be transmitted in real time to the National Agency for Medicines. It will enable National Agency for Medicines to ensure the safe use of these treatments for the pediatric population, vulnerable, and optimize monitoring in the short and long term identified or potential risks of these treatments on a developing immune system. It will also ensure the monitoring of off-label or Temporary Therapeutic Protocol / Temporary recommendation for use prescriptions and to argue recommendations for good use. For treatments whose benefit will be confirmed, these results will be useful to the medical community to define the best second-line therapeutic strategy.